CLINICAL TRIAL: NCT00507390
Title: The Effect of Omega-3 Polyunsaturated Fatty Acid Supplements on Microvolt T Wave Alternans in Patients With Ventricular Arrhythmia
Brief Title: Omega 3 Polyunsaturated Fatty Acid Supplements (PUFAs) and Microvolt T Wave Alternans (TWA) in Patients With Ventricular Arrhythmia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: funding not secured
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, AChoy, Senior Clinical Lecturer and Honorary Consultant Cardiologist, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 200306ver2
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Arrhythmia; Defibrillators, Implantable
Keywords: fish oils
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Fatty Acids, Omega-3; Omacor; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A1 (Active Comparator): n-3 PUFAs
  Interventions: Dietary Supplement: n-3 polyunsaturated fatty acids (PUFAs)
- A2 (Placebo Comparator): olive oil capsules
  Interventions: Dietary Supplement: olive oil

INTERVENTIONS:
Dietary Supplement: n-3 polyunsaturated fatty acids (PUFAs) — 2g n-3 PUFAs once daily for 8 weeks
  Other Names: Omacor
  Arms: A1
Dietary Supplement: olive oil — 1 capsule day
  Arms: A2

SUMMARY:
This is a hypothesis testing study, the hypothesis being that dietary supplements of n-PUFAs concentrates are anti-arrhythmic in ventricular arrhythmic substrates.

Study Aims: To investigate whether dietary supplements of n-3 polyunsaturated fatty acid concentrates (2g PUFAs/day, Omacor) reduces MTWA (a surrogate endpoint for ventricular arrhythmia substrate) in patients with ICDs for malignant ventricular arrhythmias.

DETAILED DESCRIPTION:
Patients from the Department of Cardiology ICD out-patient clinic, Ninewells Hospital and Medical School, will be recruited. All these patients have a history of documented ventricular arrhythmia. Data from previous studies predict that 90% of these patients will have abnormal MTWA. A total of 45 ICD patients will be recruited. The study design will be a double blind randomised placebo controlled crossover design. A baseline MTWA test will be performed and patients with an abnormal test will be selected. The patients will be randomised to receive fish oil supplements (2g/day) or placebo for 8 weeks each. At the end of each intervention period, a repeat MWTA test will be performed. A 10 ml venous blood sampled will also be collected at baseline, and after each intervention period (3 samples in total). Patients in atrial fibrillation, frequent atrial or ventricular ectopics, or with ventricular pacing from the ICD, unstable angina, NYHA IV heart failure, pregnancy or child bearing potential will be excluded from the study.

End Points of the Study. The primary endpoint will be quantitative and qualitative measures of MTWA during n-3 PUFAs treatment compared to placebo.

Statistical Analysis: Quantitative differences in MTWA measurements will be analysed by a Student's t-test and qualitative differences by a chi squared test. A probability of 0.05% will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* implantable cardiovertor defibrillators
* microvolt Twave alternans positive

Exclusion Criteria:

* unstable angina
* CHF

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change in microvolt T wave alternans status | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Allan Struthers, MD, Study Director — University of Dundee
Locations (1):
- Ninewells Hospital and medical School, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No